CLINICAL TRIAL: NCT04952220
Title: Exploratory Study of Ultrasound Signs of Native Septic Arthritis of the Knee
Acronym: USAK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-A01301-40
Record Dates: First submitted 2021-06-16; First posted 2021-07-07 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Ultrasound Therapy; Complications; Septic Arthritis; Knee Arthritis
MeSH Terms: conditions — Arthritis, Infectious | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- native septic arthritis of the knee: Describe the ultrasound abnormalities observed at D0, D10 or before surgery, 6 weeks, 3 months, 6 months, during native septic arthritis of the knee:
  thickness and vascularity of the synovial membrane, existence and measurement of joint effusion existence of articular partitioning, erosions and adjacent soft tissue involvement (muscle abscess, cellulitis)
  Interventions: Device: ultrasound

INTERVENTIONS:
Device: ultrasound — Describe the sonographic abnormalities observed at Day 0, Day 10, 6 weeks, 3 months, 6 months, during native septic arthritis of the knee

SUMMARY:
Primary objective: Description of ultrasound abnormalities seen in native septic arthritis of the knee during each visit.

Primary endpoint: Describe the ultrasound abnormalities observed on Day 0, Day 10, 6 weeks, 3 months, 6 months, during native septic arthritis of the knee.

DETAILED DESCRIPTION:
Secondary Objectives:

1. Search for poor prognostic factors in native septic arthritis of the knee.
2. To look for an association between initial sonographic factors and the use of joint lavage.
3. Look for associations between sonographic signs and clinico-radio-biologic factors at each visit (D10, 6 weeks, 3 months and 6 months)

ELIGIBILITY:
Inclusion Criteria:

* Male or female of legal age
* Bacteriologically proven native septic arthritis
* Meets the definition of septic arthritis: Bacteriological documentation of joint puncture fluid-Native articulation
* Free subject, without guardianship or trusteeship, or subordination
* Non-opposition of the patient after clear and fair information about the study

Exclusion Criteria:

* Presence of material in the affected joint
* Arthritis with Mycobacterium Tuberculosis.
* Patients benefiting from a reinforced protection, namely: minors, pregnant and/or breast-feeding women, persons deprived of liberty by a judicial or administrative decision, adults under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with native septic arthritis of the knee
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-10-27 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
description of the ultrasound abnormalities seen in native septic arthritis of the knee | Day0, Day 10 or before surgery, 6week, 3months, 6months
  Describe the ultrasonographic abnormalities seen in native septic arthritis of the knee

CONTACTS AND LOCATIONS:
Overall Officials: GERVAIS Elisabeth, Principal Investigator — Poitiers University Hospital
Locations (7):
- France (7):
  - CHU de Nantes, Nantes, Pays de la Loire Region
  - CH D'Angouleme, Angoulême
  - CH de La roche-sur-yon, La Roche-sur-Yon
  - CH De La Rochelle, La Rochelle
  - CH de Niort, Niort
  - CHU de Poitiers, Poitiers
  - CHU de Rennes, Rennes